CLINICAL TRIAL: NCT07236073
Title: The Effect of Two Different Analgesic Methods on QoR-40 Score in Primary Unilateral Knee Arthroplasties: A Prospective, Randomized Study
Brief Title: The Effect of Two Different Analgesic Methods on QoR-40 Score in Primary Unilateral Knee Arthroplasties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Principal Investigator, Ataturk University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: B.30.2.ATA.0.01.00/534
Record Dates: First submitted 2025-09-29; First posted 2025-11-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis; Knee Arthritis Osteoarthritis; Knee Arthroplasty, Total
Keywords: Osteoarthritis, Knee; Postoperative Pain
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Pain, Postoperative | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THE EFFECT OF TWO DIFFERENT ANALGESIC METHODS (Active Comparator): Patients will be randomized into two equal groups by a statistician using a computerized random numbers table:
  Group 1 (PAI+ACB): Patients will undergo periarticular injection (PAI) by the surgeon with 120 ml of local anesthetic-containing fluid before cementing, and receive an adductor canal block (ACB) with 15 ml of 0.25% bupivacaine and 1:200,000 adrenaline at the end of the operation.
  Group 2 (ACB): Patients will receive an adductor canal block catheter placed at the end of the operation and will receive 0.1% bupivacaine through this catheter as a bolus every three hours postoperatively.
  Interventions: Procedure: PRİMER TEK TARAFLI DİZ ARTOPLASTİSİNDE İKİ FARKLI ANALJEZİK YÖNTEMİ; Procedure: knee replacement

INTERVENTIONS:
Procedure: PRİMER TEK TARAFLI DİZ ARTOPLASTİSİNDE İKİ FARKLI ANALJEZİK YÖNTEMİ — PRİMER TEK TARAFLI DİZ ARTOPLASTİSİNDE İKİ FARKLI ANALJEZİK YÖNTEMİN QoR-40 PUANI ÜZERİNE ETKİSİ: PROSPEKTİF, RANDOMİZE BİR ÇALIŞMA
Procedure: knee replacement — postoperative recovery quality score

SUMMARY:
Total knee arthroplasty (TKA) is a very common operation that increases in frequency with advancing age. Similar to other surgical procedures, strategies are being developed to minimize morbidity and mortality while allowing for rapid recovery and early hospital discharge.

TKA causes moderate to severe postoperative pain for most patients. The goal of pain control after TKA is to provide excellent analgesia, early mobilization and rehabilitation, and to minimize opioid use, including overprescription of opioids after discharge Multimodal, opioid-sparing strategies for postoperative pain control include regional analgesia techniques (e.g., peripheral nerve blocks, LA infiltration, continuous epidural analgesia, neuraxial opioids) in addition to multimodal systemic analgesics.

Periarticular injection (PAI), also called local infiltration analgesia, and adductor canal block (ACB), a peripheral nerve block, are increasingly used as a component of multimodal postoperative analgesia and have been shown to reduce pain scores and opioid consumption after TKA. However, the impact of these modalities on the quality of postoperative recovery is unknown. The most widely used method of measuring this is the quality of recovery 40 (QoR 40) questionnaire. This questionnaire places increasing emphasis on measuring overall patient recovery and how quickly a patient can return to daily life after anesthesia and surgery.

Numerous studies have used the postoperative QoR-40 to compare different methods of anesthesia, adjuvants, regional analgesic techniques, and other factors on patient recovery and have been validated in Turkish.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a very common operation that increases in frequency with advancing age. Similar to other surgical procedures, strategies are being developed to minimize morbidity and mortality while allowing for rapid recovery and early hospital discharge.

TKA causes moderate to severe postoperative pain for most patients. The goal of pain control after TKA is to provide excellent analgesia, early mobilization and rehabilitation, and to minimize opioid use, including overprescription of opioids after discharge Multimodal, opioid-sparing strategies for postoperative pain control include regional analgesia techniques (e.g., peripheral nerve blocks, LA infiltration, continuous epidural analgesia, neuraxial opioids) in addition to multimodal systemic analgesics.

Periarticular injection (PAI), also called local infiltration analgesia, and adductor canal block (ACB), a peripheral nerve block, are increasingly used as a component of multimodal postoperative analgesia and have been shown to reduce pain scores and opioid consumption after TKA. However, the impact of these modalities on the quality of postoperative recovery is unknown. The most widely used method of measuring this is the quality of recovery 40 (QoR 40) questionnaire. This questionnaire places increasing emphasis on measuring overall patient recovery and how quickly a patient can return to daily life after anesthesia and surgery.

Numerous studies have used the postoperative QoR-40 to compare different methods of anesthesia, adjuvants, regional analgesic techniques, and other factors on patient recovery and have been validated in Turkish.

This study will be carried out prospectively and randomized on 60 people after obtaining the approval of the ethics committee of Atatürk University Faculty of Medicine Hospital and the written consent of the patients.

Patients will be randomized by a statistician using a computerized random numbers table and divided into 2 equal groups as Group PAI+ACB and Group ACB. All patients will undergo spinal anesthesia with 12 mg isobaric bupivacaine + 15 mcg fentanyl. Afterwards, patients in Group PAI+ACU will undergo PAI by the surgeon with a total of 120 ml of local anesthetic-containing fluid before cementing during the operation, and patients in this group will undergo ACU with 15 ml of 0.25% bupivacaine and 1:200000 thousand adrenaline at the end of the operation. Patients in group ACB will have an adductor canal block catheter placed at the end of the operation and 0.1% bupivacaine will be given postoperatively through this catheter as a bolus every three hours.

Patients will be given 1000 mg acetaminophen every six hours starting from the preoperative period, 8 mg iv dexamethasone, 4 mg iv ondansetron, 100 mcg/kg/min propofol infusion intraoperatively, 100 mcg iv fentanyl or 10 to 40 iv ketamine for analgesia when necessary, and 400 mg iboprufen every eight hours in addition to acetaminophen, 5 or 10 mg oxycodone for pain, and 25 mcg fentanyl for severe pain (VAS≥7) postoperatively. Patients will also receive 1 gram of tranexamic acid before skin incision and at the end of surgery.

QoR40 scores of the patients will be evaluated and recorded on the preoperative day and postoperative days 1 and 2 using the Turkish version of the QoR40 score.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. ASA 1-2
3. Those who gave written informed consent for their participation in the study
4. Patients undergoing unilateral primary total knee arthroplasty for end-stage osteoarthritis or rheumatoid arthritis

Exclusion Criteria:

1. Patients undergoing revision total knee arthroplasty
2. Opioid addiction
3. Preoperative hb, creatinine and electrolytes not within normal limits
4. Anticoagulants
5. Those allergic to the drugs to be used in the study
6. Those with cognitive dysfunction
7. Patients with more than 40 degrees of knee misalignment (varus or valgus)
8. Patients with advanced kidney disease (defined as GFR<30) or severe liver disease
9. Patients with poorly controlled diabetes mellitus (HbA1C>7.0 on pre-admission test)
10. BMI≥40 patients with
11. Any associated intraoperative complications
12. Pregnant or lactating female patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Levels Measured by the Visual Analog Scale (VAS) | 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 20 hours, 24 hours, 36 hours, and 48 hours after surgery.
  Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS), which ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
Quality of Recovery as Measured by the Quality of Recovery-40 (QoR-40) Questionnaire | Preoperatively (baseline), postoperative day 1, and postoperative day 2.
  The Quality of Recovery-40 (QoR-40) questionnaire will be used to evaluate patients' postoperative recovery quality. The scale ranges from 40 to 200 points, with higher scores indicating better recovery. The Turkish validated version of the QoR-40 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Dostbil, Principal Investigator — Ataturk Univercity Ethics Committee
Locations (1):
- Ataturk University, Erzurum, Erzurum, Turkey (Türkiye)